CLINICAL TRIAL: NCT07092267
Title: A Multiple Center, Prospective, Single-arm, Open Label, Pilot Study to Evaluate the Safety and Efficacy of ArtiFix® Sealant Graft in Subjects Requiring Dural Repair Following Neurosurgery
Brief Title: Safety and Efficacy Evaluation of ArtiFix® Sealant Graft in Subjects Requiring Dural Repair Following Neurosurgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nurami Medical Ltd (Other)
Collaborators: KCRI (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-02-1026
Record Dates: First submitted 2025-07-01; First posted 2025-07-29 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Cerebrospinal Fluid Leak; Dural Tear
MeSH Terms: conditions — Cerebrospinal Fluid Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects requiring Dural repair during elective neurosurgery procedures. (Experimental): Men and women scheduled for an elective cranial or spinal surgery that requires Dural repair during elective neurosurgery procedure. The investigated device is a surgical Dural sealant graft intended to close Dural defects.
  Interventions: Device: ArtiFix® is a surgical dural sealant graft intended to close dural defects following cranial and spine surgeries.

INTERVENTIONS:
Device: ArtiFix® is a surgical dural sealant graft intended to close dural defects following cranial and spine surgeries. — ArtiFix® is a synthetic surgical dural sealant graft intended to close dural defects following cranial and spine surgeries. ArtiFix® adheres to the dura, so that sutures are not required to prevent cerebrospinal fluid (CSF) leakage.

SUMMARY:
The purpose of this clinical study is to evaluate and establish the safety and efficacy of the ArtiFix® device in subjects scheduled for cranial or spinal surgery that requires Dural repair (membrane that covers the brain and spinal cord). The investigated device will be implanted during the neurosurgical procedure and participants will be evaluated at 30, 120 and 330 days after the procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject between the ages of 22-65 (inclusive)
2. Subject is scheduled for an elective cranial or spinal surgery with a single dural defect that could not be completely repaired by primary suture. The dural defect must not exceed 6cm2 (e.g. defects of sizes 2cm X 3cm, 1cm X 5cm, can be included). The defect can be completely repaired/closed by a dural sealant graft with an overlap of 6 mm with the surrounding intact dura (only 1 graft can be implanted in each subject in a single location).
3. Subject has undergone imaging (such as, CT or MRI) in the past 6 months before enrolment.
4. Surgical wound is expected to be Class I/clean.
5. Subject understands the study requirements and procedures, can provide written Informed Consent and is able and willing to adhere to the required follow-up visits and testing.

Exclusion Criteria:

1. Subject has known hydrocephalus.
2. Subject is unable to undergo MRI after the surgery.
3. Subject's life expectancy is less than 12 months.
4. Significant intraoperative hemorrhage that mandates blood transfusion.
5. Subject has a local or systemic infection (e.g. urinary tract infection (UTI), active pneumonia etc.) or evidence of any surgical site infection, fever > 38.3°C, positive blood culture and/or a positive chest x-ray for acute inflammatory process.
6. Subject has acquired or congenital compromised immune system and/or autoimmune disease, and/or is taking chronic immunosuppressant agents at baseline.
7. Subject will require use of other forms of dural repair (i.e. dural graft or sealant).
8. Subject is intended to undergo craniectomy wherein bone flap will not be returned.
9. Subject with a compromised wound healing process due to past treatments (e.g. chemotherapy, radiation therapy, severe diabetes etc.) or other concurrent conditions (e.g. long-standing steroids treatment).
10. Subject has been clinically diagnosed with malignancy (other than basal cell carcinoma or low-grade glioma), uncontrolled diabetes (A1C>6.5%), sepsis, and systemic collagen disease.
11. Subject had chemotherapy and/or radiotherapy in the past 12 weeks before surgery or is planned to have chemotherapy or radiotherapy less than 12 weeks after surgery.
12. Subject is an acute cranial trauma surgical case or had intracranial hemorrhage from any cause (hemorrhagic stroke, ruptured aneurysm etc.).
13. Subject that has a concurrent disease or symptoms or conditions that would place the patient in excessive risk to the planned surgery - defined by PI.
14. Subject had a previous neurosurgery in the same anatomical site.
15. Subject was diagnosed with clinically significant coagulopathy as determined by the surgeon.
16. Subject is participating in another clinical trial using investigational devices/drugs
17. Subjects who previously participated in any investigational drug or device study within 30 days of screening
18. Subject has known history of sensitivity or allergy to any component of the ArtiFix®.
19. Female subjects who are breastfeeding, pregnant or interested in becoming pregnant during the duration of the study.
20. Any condition or abnormality which in the opinion of the investigator may jeopardize the subject's safe participation.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of CSF leakage rate up to 120 days after ArtiFix® implantation. | up to 120 days after ArtiFix® implantation

SECONDARY OUTCOMES:
Evaluation of CSF leakage rate via MRI at 120 days after ArtiFix® implantation Evaluation of CSF leakage rate via MRI at 330 days after ArtiFix® implantation | at 120 and 330 days after ArtiFix® implantation.
To evaluate the frequency and severity of device-related adverse events, up to 330 days post ArtiFix® implantation. | up to 330 days post ArtiFix® implantation.
Wound healing at implant site up to 30 days after implantation. | Up to 30 days after implantation.
Device Handling Characteristics, as reported by the surgeon [e.g. Ease of Use, Strength, Seal Quality, Reapplication (if occurred), adhesion to surgical tools]. Device Handling Characteristics reported by user experience questionnaire. | Following investigational device implantation on the day of the surgical procedure.
Magnetic Resonance Imaging at the 120 and 330 days follow-up, to determine the presence or absence of the following conditions: • Adhesion formation • Scarring • Brain edema adjacent to device implant site | At the 120 and 330 days follow-up visits

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Milbaum, Study Director

IPD SHARING:
Plan to Share IPD: Undecided